CLINICAL TRIAL: NCT05347550
Title: Examining the Benefit of Graduated Compression Stockings in the Prevention of vEnous Thromboembolism in Low-risk Surgical Patients: a Multicentre Cluster Randomised Controlled Trial (PETS)
Brief Title: Examining the Benefit of Graduated Compression Stockings in the Prevention of vEnous Thromboembolism in Low-risk Surgical Patients
Acronym: PETS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Edinburgh (Other); Universidad de Granada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22CX7651
Record Dates: First submitted 2022-04-08; First posted 2022-04-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism
Keywords: Cluster; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - No graduated compression stockings (No Intervention): In those centres randomised to the control arm, participants will not receive Graduated Compression Stockings (GCS).
- Intervention - The provision of graduated compression stockings (Experimental): Centres randomised to the intervention arm, which is the current standard of care, will consist of participants receiving Graduated Compression Stockings (GCS). Clinical staff (e.g. theatre support workers) will issue stockings to all patients who are scheduled to undergo short-stay surgery. Participants will be instructed to wear their stockings just before undergoing the surgical procedure and to remove the stockings as soon as they are ambulant (i.e. after the procedure).
  Interventions: Other: Graduated Compression Stockings - Thromboembolic deterrent stockings

INTERVENTIONS:
Other: Graduated Compression Stockings - Thromboembolic deterrent stockings — Centres randomised to the intervention arm will consist of participants receiving GCS.
  Arms: Intervention - The provision of graduated compression stockings

SUMMARY:
Hospital acquired thrombosis describes blood clots that form in the legs and lungs after someone is treated in hospital. Clots in the leg can cause swelling, pain and other problems. If a clot in the leg travels to the lungs, it may be life threatening. Having surgery increases the risk of developing blood clots.

People having short-stay surgery (who either go home the same day or who stay overnight but go home shortly afterwards) are at a much lower risk of developing a blood clot than those who stay in hospital for longer. These low-risk people are often given elastic stockings (which squeeze the leg muscles) to reduce the chance of a blood clot.

The risks of wearing the stockings are low but they can be uncomfortable. In the UK, there are over a million short stay surgeries performed each year and most of these people are given elastic stockings to wear. Stockings cost the NHS a lot of money and it remains unknown if they work.

This study will investigate if it is worthwhile to continue using elastic stockings in people having surgery where the risk of developing blood clots is low. Adults (over 18-years) who are at low risk of developing blood clots (assessed using a nationally recognised tool) will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-59 years of age) scheduled to undergo a surgical procedure with a hospital stay <48 hours
* Individuals assessed as being at low-risk of developing VTE as per the DHRA Tool (i.e. no assessed thrombosis risk factors / scoring 0)

Exclusion Criteria:

* Individuals with a contraindication to GCS
* Individuals assessed as being at moderate or high-risk of VTE as per the DHRA tool
* Individuals requiring therapeutic anticoagulation
* Individuals with thrombophilia/ thrombogenic disorder
* Individuals with a previous history of VTE
* Individuals requiring intermittent pneumatic compression therapy beyond theatre and recovery
* Individuals requiring extended thromboprophylaxis beyond discharge
* Female patients of childbearing age who have a positive pregnancy test
* Individuals with lower limb immobilisation
* Inability to provide informed consent

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21472 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of symptomatic VTE within 90 days | 90-days
  The rate of symptomatic VTE for surgical patients undergoing short-stay procedures assessed as being at low-risk of VTE

SECONDARY OUTCOMES:
Mortality | 90-days
Quality of Life | 7 and 90-days
  Quality of Life assessed using the EQ-5D
Adverse events related to GCS | 7-days
  Adverse events related to GCS for those in the intervention arm only
Health Economic Outcome | 2 years
  Incremental Cost-Effectiveness Ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London
Locations (9):
- United Kingdom (9):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Frimley Health NHS Foundation Trust, Camberley
  - Queen Victoria Hospital NHS Foundation Trust, East Grinstead
  - Imperial College Hospital NHS Foundation Trust, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Sherwood Forest Hospital NHS Foundation Trust, Nottingham
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: No